CLINICAL TRIAL: NCT01198340
Title: Evaluation of Optimal Dose of Local Anesthetics for Patient Controlled Continuous Femoral Nerve Block With Sciatic Nerve Block After Total Knee Arthroplasty
Brief Title: Evaluation of Optimal Dose of Local Anesthetics for Patient Controlled Continuous Femoral Nerve Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Okayama University (Other)
Responsible Party: Hideki Taninishi, Okayama University Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TKAFEMORAL-2010; UMIN000004155 (Registry Identifier: UMIN.JP)
Record Dates: First submitted 2010-09-08; First posted 2010-09-10 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2010-08

CONDITIONS: Arthropathy of Knee Joint

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- With basal local anesthetics (Active Comparator)
  Interventions: Procedure: PC-FNB with basal administration of local anesthetics
- Without basal local anesthetics (Experimental)
  Interventions: Procedure: PC-FNB without basal local anesthetics

INTERVENTIONS:
Procedure: PC-FNB with basal administration of local anesthetics — Administration of 0.2% ropivacaine for femoral nerve block with 3 ml/h of basal dose, 5ml bolus by the patient, 60 minutes of lock out time.
  Other Names: PC-FNB with basal ropivacaine administration
  Arms: With basal local anesthetics
Procedure: PC-FNB without basal local anesthetics — Administration of 0.2% ropivacaine for femoral nerve block without basal dose, with 8 ml bolus by the patient, 60 minutes of lockout time.
  Other Names: PC-FAB without basal ropivacaine administration
  Arms: Without basal local anesthetics

SUMMARY:
To evaluate an analgesic effect without basal administration of local anesthetics for patient-controlled femoral nerve block (with sciatic nerve block) after total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 20 yrs old scheduled for total knee arthroplasty

Exclusion Criteria:

* none

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-03 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
pain scores by use of numerous rating scale (NRS) | 4 days after the surgery

SECONDARY OUTCOMES:
dose of local anesthetics | 4 days after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hideki Taninishi, MD, PhD, Principal Investigator — Okayama University
Locations (1):
- Anesthesiology and Resuscitology, Okayama University Hospital, Okayama, Okayama-ken, Japan